CLINICAL TRIAL: NCT00484913
Title: Effects of Abdominal Hot Compresses on Indocyanine Green Elimination - a Randomized Cross Over Study in Healthy Subjects
Brief Title: Effects of Abdominal Hot Compresses on Indocyanine Green Elimination in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: LW05
Record Dates: First submitted 2007-06-08; First posted 2007-06-12 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
Keywords: healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: abdominal hot compress

SUMMARY:
We investigated, whether abdominal hot compresses effect hepatic blood flow. Our hypothesis was, that the hot compresses might either by local vasomotor-reflex or by decreasing the tone of the sympathetic nerve system increase hepatic blood flow.

DETAILED DESCRIPTION:
Abdominal hot compresses are traditionally used by patients with liver diseases as self help. This study investigated the effect of abdominal hot compresses on hepatic blood flow measured by elimination of indocyanine green (ICG), a non-toxic green dye. It was presumed, that abdominal hot compresses increase hepatic blood flow either by local vasomotor-reflex or by decreasing the tone of the sympathetic nerve system.

In healthy volunteers ICG elimination was measured with and without hot compress at two investigations in a weekly interval. At each investigation ICG was injected as bolus after a rest period of 10 minutes. After the injection blood was taken in regular intervals for analysis of ICG concentration over a period of 40 minutes and half life was calculated.

The time interval between the investigations was 8 days, the sequence was randomly assigned.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* iodine allergy
* any acute or chronic disease [with exception of pollinosis because it is common]
* elevated levels of alanine amino transferase [ALT], aspartate amino transferase [AST], gamma glutamyltransferase [GGT] or bilirubin
* heat urticaria
* pregnancy
* alcohol intake >30 g/d
* any medication except contraceptives
* body mass index (BMI) >30 kg/m2

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2003-09; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Indocyanine green half life | 40 minutes

SECONDARY OUTCOMES:
heart rate, blood pressure | 40 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Roman Huber, Dr., Principal Investigator — Department of Internal Medicine II, Freiburg University Hospital, Germany
Locations (1):
- Department of Internal Medicine II, Freiburg University Hospital, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Huber R, Weisser S, Luedtke R. Effects of abdominal hot compresses on indocyanine green elimination--a randomized cross over study in healthy subjects. BMC Gastroenterol. 2007 Jul 10;7:27. doi: 10.1186/1471-230X-7-27. PMID 17623067